CLINICAL TRIAL: NCT04509713
Title: Using Medical-detection Dogs to Identify People With SARS-CoV-: Phase I: Proof-of-concept Studies
Brief Title: Canine COVID-19 Detection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ARCTEC (Industry)
Collaborators: Durham University (Other); Cardiff University (Other); Medical Detection Dogs (Unknown)
Responsible Party: Sponsor
Other Study IDs: LSH1285
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- infected/positive group: asymptomatic or mildly symptomatic participants positive for SARS-CoV-2 RNA
  Interventions: Behavioral: Collection of odour samples
- uninfected/negative group: no evidence of SARS-CoV-2 by real-time RT-PCR
  Interventions: Behavioral: Collection of odour samples

INTERVENTIONS:
Behavioral: Collection of odour samples — Samples of breath odours will be passively collected while participants wear the mask while breathing naturally, for at least 3 h. Skin odours will be passively collected by participants wearing the shirt and nylon socks for at least 12 h.

SUMMARY:
Dogs are some of nature's greatest detectives, owing to their incredible sense of smell and ability to be trained. Most of us will be familiar with seeing trained sniffer dogs at airports looking for drugs and other prohibited items, but their skills don't stop there. The use of medical detection dogs is becoming increasingly common, as they are able to identify cancers, changes in blood sugar levels and even predict seizures. These are just a few examples of dogs playing a key role in public health. Many diseases can alter the way humans smell. A study undertaken by the London School of Hygiene & Tropical Medicine (LSHTM) and Durham University has shown that dogs are able to accurately diagnose malaria. The investigators know that respiratory illnesses can alter your body odours, and thus the investigators plan to determine whether dogs are able to identify the novel coronavirus known as COVID-19 (or SARS-CoV-2).

COVID-19 can present itself asymptomatically (i.e. causing no apparent symptoms), which could lead to the spread of infection in the population. The investigators believe that dogs may be able to identify asymptomatic patients, as well as those who have mild symptoms (symptoms not requiring treatment, hospital stay or limiting normal activities). It is thought that a single medical detection dog stationed within an airport would be able to screen up to 750 people for COVID-19 infection in just 1 hour, informing those who are infected to isolate, preventing further spread of the disease.

In order to determine whether it is possible for dogs to accurately diagnose COVID-19, the investigators must first collect samples. NHS staff and members of their households that are eligible for SARS-CoV-2 screening, have been selected to participate in this study due to their potential exposure to this disease agent. In addition, participants from the general population who are displaying mild COVID-19 symptoms or have been exposed to COVID-19 will be recruited via hospitals, testing centers, outbreak testing programs and home testing programs. Initially, participants will attend their screening test as planned or confirm that they have had a swab test within the previous 24 hours. Immediately following this, the investigators will ask participants to collect samples of breath odour and body odour, which will be collected passively through the wearing of face masks, shirts, and nylon socks. The investigators will ask to be provided with the results of the SARS-CoV-2 screening swab, which will allow for us to determine whether participants are positive or negative for SARS-CoV-2. These odour samples will be grouped by positive or negative test results, and transported to LSHTM where these will be processed in order to prevent contact with the virus, negating the risk for dogs and their handlers.

A pilot study will be undertaken to confirm whether dogs are able to distinguish between positive and negative samples using traditional sniffer dog training methods. If this is possible, the investigators will proceed to the main study to determine the accuracy (known as sensitivity and specificity) of the dogs' ability to identify the virus. Both the handler and the dogs themselves will be 'blinded' to the samples, and thus unaware of which sample is which. When the data generated by these tests is entered, it will be confirmed whether or not the samples have been correctly identified.

The dogs will be trained to detect and report the detection of the volatile odours characteristic of COVID-19 infection. For quality control purposes the investigators also aim to characterise the COVID-19 odour profile by analysing samples with a special process called GC (gas chromatography) and/or GC-MS (gas chromatography coupled mass spectrometry). This will help to inform the identification of compounds showing differences between infected and non-infected samples.

The investigators believe that this work could be useful in the fight against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Due to have a coronavirus swab test or have had a swab test conducted in the previous 24 hours
* Aged ≥ 16 years
* Have suspected mild COVID-19 symptoms or have been exposed to COVID-19, or are NHS staff or household member of NHS staff
* No evidence of previous laboratory confirmed SARS-CoV-2
* Written informed consent provided
* Willing and able to wear a face mask for at least 3h
* Willing and able to wear nylon socks for at least 12 h
* Willing and able to wear a shirt for at least 12 h
* Willing and able to provide a copy of their coronavirus swab test result

Exclusion Criteria:

* Aged < 16 years
* Evidence of moderate to severe illness with symptoms compatible with SARS-CoV-2 infection which require hospital admission
* Previous (>24 hours) clinical diagnosis of COVID-19
* Previous (>24 hours) laboratory confirmed SARS-CoV-2 infection
* Written informed consent not provided
* Unable or unwilling to wear a facemask for at least 3 h
* Unwilling or unable to wear nylon socks for at least 12 h
* Unwilling or unable to wear a shirt for at least 12 h
* Unwilling or unable to provide a copy of their coronavirus swab test result

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Have suspected mild COVID-19 symptoms or have been exposed to COVID-19, or are NHS staff or household member of NHS staff
Sampling Method: Non-Probability Sample
Enrollment: 16250 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity precision of dogs to detect people with COVID-19 by their odour. | 4 months
  The main study is designed to measure the sensitivity and specificity of the dogs to detect participants infected with SARS-CoV-2. Dogs will be trained for a period of 6-8 weeks to give a behavior response to positive samples. During training the reaction of each dog to a positive sample will be observed (i.e. standing, sitting or lying down) and this indicating behaviour reinforced by rewarding the dog. The dog's diagnostic accuracy will then be determined in a double-blinded study. Here the trainer and technician using the computer to record the results of the study are blinded to the identity of each sample until the trainer calls the final decision (positive or negative) based on the response of the dog to the sample.

SECONDARY OUTCOMES:
Identification of the volatile profile that is specific to asymptomatic or mild symptomatic participants with SARS-CoV-2 compared with uninfected individuals. | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- ARCTEC, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guest C, Dewhirst SY, Lindsay SW, Allen DJ, Aziz S, Baerenbold O, Bradley J, Chabildas U, Chen-Hussey V, Clifford S, Cottis L, Dennehy J, Foley E, Gezan SA, Gibson T, Greaves CK, Kleinschmidt I, Lambert S, Last A, Morant S, Parker JEA, Pickett J, Quilty BJ, Rooney A, Shah M, Somerville M, Squires C, Walker M, Logan JG; COVID Dogs Research Team. Using trained dogs and organic semi-conducting sensors to identify asymptomatic and mild SARS-CoV-2 infections: an observational study. J Travel Med. 2022 May 31;29(3):taac043. doi: 10.1093/jtm/taac043. PMID 35325195